CLINICAL TRIAL: NCT05968430
Title: An Open-Label Extension Study to Assess the Long-Term Safety, Efficacy, and Tolerability of Lorundrostat in Subjects With Hypertension
Brief Title: Open-Label Extension (OLE) Study to Assess Safety, Efficacy, and Tolerability of Lorundrostat in Subjects With Hypertension
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Mineralys Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MLS-101-901
Record Dates: First submitted 2023-07-14; First posted 2023-08-01 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2025-06

CONDITIONS: Hypertension
Keywords: Blood pressure; Uncontrolled hypertension; Hypertension; Hypertensive
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Masking Description: Eligible subjects participating in the RTW will receive double-blind treatment with matching placebo. Upon completion, subjects will return to open-label treatment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Open-Label Arm (Experimental): lorundrostat once daily for 52 weeks depending on when the subject enrolled
  Interventions: Drug: lorundrostat
- RTW Substudy (Experimental): lorundrostat or placebo once daily for 4 weeks starting at week 12, in the double-blind randomized treatment withdrawal substudy
  Optional for subjects from the MLS-101-301 parent study only
  Interventions: Drug: lorundrostat; Drug: Placebo
- Optional Continuation Period (Experimental): lorundrostat once daily from week 52 or until marketing authorization or early termination of the trial by the sponsor
  Interventions: Drug: lorundrostat

INTERVENTIONS:
Drug: lorundrostat — Tablet, administered orally
Drug: Placebo — Tablet, administered orally
  Arms: RTW Substudy

SUMMARY:
This study is to evaluate the long-term safety, efficacy and tolerability of lorundrostat (an aldosterone synthase inhibitor) in subjects with hypertension

DETAILED DESCRIPTION:
The purpose of the study is to evaluate the long-term safety, efficacy, and tolerability of lorundrostat (an aldosterone synthase inhibitor) in subjects with hypertension.

This study consists of an open label treatment period of 52 weeks followed by a 2-week safety follow-up period. Eligible subjects for MLS-101-901 are those who were enrolled in one of the eligible parent studies, meet the eligibility criteria for this protocol, and agree, by signing an informed consent form (ICF), to transition to this open label extension (OLE) study at either the end-of-study (EoS) visit or the end-of-treatment (EoT) visit as required in the parent study protocol.

A Randomized Treatment Withdrawal (RTW) substudy will be performed in a subset of subjects meeting eligibility criteria.

Subjects who complete the open label treatment period will be invited to consent to an optional continuation period where they may remain on study until marketing authorization or early termination of the trial by the sponsor.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent signed by the participant, obtained before any study-related assessment is performed
2. At least 18 years of age at the time of signing the informed consent form (ICF)
3. Completed the EoT or EoS Visit (as applicable) in a lorundrostat study with the option of transitioning to the OLE study, in accordance with the parent study protocol
4. Fertile male subjects and female subjects of childbearing potential, and their partners, must agree to use an acceptable method of contraception from study entry to 28 days after the last dose of study drug
5. Willing and able to comply with the study instructions and attend all scheduled study visits

   [Randomized treatment withdrawal substudy only]
6. Written informed consent to participate in the RTW substudy signed by the participant, obtained before any RTW study-related assessment is performed

Exclusion Criteria:

1. Women who are pregnant, plan to become pregnant, or are breast-feeding
2. Use, or anticipated use during the course of the study, of a prohibited medication as listed in Section 6.7.1 of the protocol
3. In the opinion of the Investigator, any condition that will preclude participation in the study

   [Randomized treatment withdrawal substudy only]
4. Non-compliance with study medication(s) (defined as taking <75% or >125% of the study drug provided) during the first 12 weeks of MLS-101-901

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1076 (Actual)
Dates: Start 2023-07-14 (Actual); Primary Completion 2025-12-30 (Actual); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change from MLS-101-301 baseline automated office blood pressure | Week 36
  Change from MLS-101-301 baseline automated office blood pressure (AOBP) systolic blood pressure (SBP) at MLS-101-901 Week 36 in subjects who were enrolled in the lorundrostat arms of MLS-101-301 and were not assigned to the placebo arm of the MLS-101-901 RTW substudy
Change at MLS-101-901 Week 16 (RTW Week 4) from MLS 101-901 Week 12 (RTW substudy baseline) in AOBP SBP in subjects enrolled in RTW | Week 16

CONTACTS AND LOCATIONS:
Locations (177):
- United States (128):
  - Accel Research Sites (ARS) - Birmingham Clinical Research Unit, Birmingham, Alabama
  - G & L Research LLC, Foley, Alabama
  - Chandler Clinical Trials, Chandler, Arizona
  - Arizona Kidney, Glendale, Arizona
  - AKDHC Medical Research Services, AZ, Phoenix, Arizona
  - Noble Clinical Research, Tucson, Arizona
  - Del Sol Research Management, LLC, Tucson, Arizona
  - Entertainment Medical Group, Inc, Beverly Hills, California
  - CA Institute of Renal Research, CA, Chula Vista, California
  - Amicis Research Center - Vacaville, Fairfield, California
  - Amicis Research Center - Granada Hills, Granada Hills, California
  - Marvel Clinical Research 002, LLC, Huntington Beach, California
  - University of California San Diego (UCSD) - Altman Clinical and Translational Research Institute (ACTRI), La Jolla, California
  - Clinical Trials Research (CTR) - Lincoln, Lincoln, California
  - Academic Medical Research Institute (AMRI) - Los Angeles, Los Angeles, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Amicis Research Center - Mission Hills, Northridge, California
  - Amicis Research Center-Northridge, Northridge, California
  - Northridge Clinical Trials, Northridge, California
  - Pasadena Clinical Trials, Pasadena, California
  - Empire Clinical Research, Pomona, California
  - Clinical Trials Research (CTR) - Sacramento, Sacramento, California
  - Triwest Research Associates, San Diego, California
  - San Jose Clinical Trials, San Jose, California
  - Amicis Research Center - Valencia, Valencia, California
  - Kidney & Hypertension Center - Victorville, Victorville, California
  - Blue Coast Research Center (BCRC), Vista, California
  - Accelerated Enrollment Solutions (AES) -Vista/Synexus (Radiant Research), Vista, California
  - Colorado Kidney (Denver) Nephrology, Denver, Colorado
  - CMR of Greater New Haven, Hamden, Connecticut
  - Qway Research, Hialeah, Florida
  - Indago Research and Health Center, Hialeah, Florida
  - Clinical Neuroscience Solutions, Inc, Jacksonville, Florida
  - Nuovida Research Center Corp, Miami, Florida
  - Clinical Neuroscience Solutions, Inc, Orlando, Florida
  - Nephrology Associates of Central Florida, Orlando, Florida
  - AES - Orlando, Orlando, Florida
  - Pines Care Research Center, Pembroke Pines, Florida
  - Patron Medical - Andres Patron D.O. (Patron Ventures, LLC), Pembroke Pines, Florida
  - Progressive Medical Research, Port Orange, Florida
  - Infigo Clinical Research (Mid Florida), Sanford, Florida
  - Clinical Research of West Florida, Inc., Tampa, Florida
  - AES The Villages, The Villages, Florida
  - Palm Beach Diabetes and Endocrine Specialists, PA (PBDES) - West Palm Beach Office), West Palm Beach, Florida
  - American Clinical Trials, Acworth, Georgia
  - Morehouse School of Medicine, Atlanta, Georgia
  - Coastal Medical, Brunswick, Georgia
  - Accel Research Sites, Decatur, Georgia
  - Georgia Clinical Research, LLC, Lawrenceville, Georgia
  - Alta Pharmaceutical Research Center, Peachtree Corners, Georgia
  - Elite Clinical Trials, Blackfoot, Idaho
  - Meridian Family Medicine, Meridian, Idaho
  - AES Chicago/Synexus Clinical Research, Chicago, Illinois
  - Eagle Clinical Research, Chicago, Illinois
  - The University of Chicago Medicine, Chicago, Illinois
  - Healthcare Research Network - Chicago, Flossmoor, Illinois
  - Koch Family Medicine, S.C, Morton, Illinois
  - Southern Illinois School of Medicine, Springfield, Illinois
  - Hendricks Regional Health Medical Group - Lizton Family Medicine, Brownsburg, Indiana
  - AES Evansville/Synexus Clinical Research, Evansville, Indiana
  - ASHA Clinical Research- Munster, LLC, Hammond, Indiana
  - The Research Group of Lexington, LLC, Lexington, Kentucky
  - Nephrology Associates of Kentuckiana, Louisville, Kentucky
  - Alliance for Multispecialty Research, LLC, New Orleans, Louisiana
  - Northwest Louisiana Nephrology, LLC - Shreveport, Shreveport, Louisiana
  - Boston Clinical Trials, Boston, Massachusetts
  - ActiveMed Practices & Research LLC, Methuen, Massachusetts
  - Hattiesburg Clinic, Petal, Mississippi
  - Healthcare Research Network-Hazelwood, Hazelwood, Missouri
  - Clinical Research Consultants (CRC) - Kansas City, Kansas City, Missouri
  - Quality Clinical Research, Omaha, Nebraska
  - Henderson Clinical Trials, Henderson, Nevada
  - Synexus Clinical Research US, Inc., Henderson, Nevada
  - Sierra Clinical Research, Las Vegas, Nevada
  - Oasis Clinical Trials, Las Vegas, Nevada
  - Las Vegas Clinical Trials, North Las Vegas, Nevada
  - Renown Regional Medical Center, Reno, Nevada
  - Albany Medical College, Albany, New York
  - Erie County Medical Center, Buffalo, New York
  - AES New York/Synexus Clinical Research, New York, New York
  - Columbia University, New York, New York
  - Triad Internal Medicine, Asheboro, North Carolina
  - East Carolina University (ECU) Physicians - East Carolina Heart Institute - East Carolina University Location, Greenville, North Carolina
  - Physician's East Endocrinology, Greenville, North Carolina
  - Carteret Medical Group, Morehead City, North Carolina
  - Lucas Research, New Bern, North Carolina
  - Research Innovations (Elligo Health Research), Beavercreek, Ohio
  - Diabetes & Endocrinology Associates of Stark County, Canton, Ohio
  - Intrepid Research, Cincinnati, Ohio
  - Cleveland Clinic - Main Campus, Cleveland, Ohio
  - Arthritis & Osteoarthritis Center of SW Ohio/ dba STAT Research, Vandalia, Ohio
  - Lynn Institute of Norman (LION Research), Norman, Oklahoma
  - Willamette Valley Clinical Studies, Eugene, Oregon
  - AMS Cardiology (Elligo), Horsham, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Preferred Primary Care Physicians, Pittsburgh, Pennsylvania
  - Accelerated Enrollment Solutions (AES) - Anderson, Anderson, South Carolina
  - Wake Research - Notus Clinical Trials, LLC, Charleston, South Carolina
  - Coastal Carolina Research Center, North Charleston, South Carolina
  - Chattanooga Medical Research, Chattanooga, Tennessee
  - AMR - Knoxville, Knoxville, Tennessee
  - Clinical Neuroscience Solutions, Inc, Memphis, Tennessee
  - Lifedoc Research, Memphis, Tennessee
  - Vanderbilt University Medical Center (VUMC), Nashville, Tennessee
  - Punzi Medical Center, Carrollton, Texas
  - AES - Dallas Fort Worth, Dallas, Texas
  - David Turbay, MD, PLLC (Elligo Health Research), El Paso, Texas
  - Synergy Groups Medical - Bissonet Site, Houston, Texas
  - Juno Research, LLC, Houston, Texas
  - Gulf Coast Clinical Research, Houston, Texas
  - Medical Colleagues of Texas, LLP (Elligo Health Research), Katy, Texas
  - R & H Clinical Research, Katy, Texas
  - Gamma Medical Research, Inc, McAllen, Texas
  - Office of Audrey L. Jones, DO, McAllen, Texas
  - PRX Research - Mesquite, Mesquite, Texas
  - Synergy Groups Medical - Missouri City, Missouri City, Texas
  - ACRC Trials - Legacy Medical Village Location, Plano, Texas
  - Clinical Investigations of Texas (CIT), Plano, Texas
  - ACRC Trials - Legacy Medical Village, Plano, Texas
  - Sun Research Institute (SRI) - San Antonio, San Antonio, Texas
  - San Antonio ClinicalTrials, San Antonio, Texas
  - Discovery Clinical Trials, San Antonio, Texas
  - Sugar Lakes Family Practice (Elligo Health Research), Sugar Land, Texas
  - The University of Utah, Salt Lake City, Utah
  - Velocity Clinical Research, West Jordan, Utah
  - Burke Internal Medicine, Burke, Virginia
  - Eastern VA Medical School, Norfolk, Virginia
  - Office of Ramon Mendez, Woodbridge, Virginia
- Australia (5):
  - Renal Research - Gosford, Gosford, New South Wales
  - Castle Hill Medical Centre, Castle Hill
  - The University of Western Australia - School of Medicine and Pharmacology - Royal Perth Hospital Unit., Perth
  - University of Sunshine Coast Clinical Trial Centre, Sippy Downs
  - AusTrials - Taringa, Taringa
- Bulgaria (5):
  - Medical Center New Polyclinic Gabrovo Ltd., Gabrovo
  - Medical Center, Pleven
  - Medical Center Hera EOOD - Sofia, Sofia
  - ASOMHIDC - Individual practice Cardio Tonus EOOD, Sofia
  - DCC 1 - Veliko Tarnovo" EOOD, Veliko Tarnovo
- Centre Medical L'Acadie - Montreal, Montreal, Quebec, Canada
- Centre Hospitalier Annecy Genevois - Site d'Annecy, Annecy, France
- Germany (5):
  - FutureMeds GmbH, Berlin
  - MVZ Jung GbR, Deggingen
  - Klinische Forschung Dresden GmbH, Dresden
  - Uniklinik Leipzig, Klinik und Poliklinik für Kardiologie, Leipzig
  - Herzzentrum Leipzig, Leipzig
- Italy (6):
  - IRCCS AOU di Bologna - Policlinico S. Orsola, Bologna
  - Azienda Ospedaliero-Universitaria di Ferrara - Arcispedale Sant'Anna, Ferrara
  - IRCCS Ospedale Policlinico San Martino, Genova
  - University of Messina, Messina
  - Azienda Ospedaliero Universitaria Pisana, Pisa
  - University of Rome Sapienza, AO Sant'Andrea, Roma
- Amsterdam AMC, Amsterdam, Netherlands
- Poland (6):
  - Samodzielny Publiczny Szpital Kliniczny im. Andrzeja Mielęckiego (SPSKM), Katowice
  - Futuremeds Lodz, Lodz
  - Futuremeds Olsztyn, Olsztyn
  - Etyka Osrodek Badan Klinicznych, Olsztyn
  - Clinmedica Research, Skierniewice
  - ETG Warszawa, Warsaw
- Latin Clinical Trial Center, San Juan, Puerto Rico
- Romania (5):
  - Centrul Medical Unirea SRL Brasov (Regina Maria), Brasov
  - Delta Health Care SRL Bucuresti - Spitalul Academic Ponderas (Regina Maria), Bucharest
  - Spitalul Clinic Judetean de Urgenta Targu Mures, Târgu Mureş
  - MEDICALI'S SRL Timisoara, Timișoara
  - Spitalul Clinic Judetean de Urgenta "Pius Branzeu" Timisoara, Timișoara
- Spain (4):
  - Complejo Hospitalario Universitario de Badajoz (CHUB) (Hospital Infanta Cristina), Badajoz
  - Hospital Universitario Reina Sofia, Córdoba
  - Hospital Universitario Virgen de las Nieves, Granada
  - Hospital Clínico Universitario Valencia, Valencia
- United Kingdom (9):
  - Newquay Health Centre, Newquay, Cornwall
  - Fowey River Practice, Fowey, England
  - Queen Elizabeth University Hospital, Glasgow, Scotland
  - Rowden Surgery Rowden Medical Partnership, Chippenham, Wilts
  - Cambridge University Hospitals NHS Foundation Trust, Cambridge
  - Epsom and St Helier University Hospitals NHS Trust, Carshalton
  - Barts Health Nhs Trust, London
  - Knowle House Surgery, Plymouth
  - Rame Medical Limited, Torpoint